CLINICAL TRIAL: NCT06647160
Title: Safety and Efficacy of Blue Star MAX-5 Lenses in Mvopia Control: A Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy of Blue Star MAX-5 Lenses in Myopia Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024KYPJ115
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Myopia, Progressive
Keywords: concentric columnar microstructure; Myopia control
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Blue star MAX-5 spectacle lens
  Interventions: Device: Blue star MAX-5 spectacle lens
- Control (Active Comparator): Single-vision spectacle lens
  Interventions: Device: Single-vision spectacle lens

INTERVENTIONS:
Device: Blue star MAX-5 spectacle lens — The children in the experimental group will wear Blue star MAX-5 spectacle lens and receive follow-up examinations every half year.
  Arms: Intervention
Device: Single-vision spectacle lens — The children in the single-vision lenses group will wear single-vision spectacle lens and receive follow-up examinations every half year.
  Arms: Control

SUMMARY:
The goal of this randomised controlled clinical trial is to compare the effects of a new type of concentric columnar microstructure lens and single-vision spectacle lenses on myopia progression in Chinese children aged 8-11 years with refractive error ranging from -0.50D to -6.00D. Participants will wear spectacles and receive follow-up examinations every half year.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8 to 11 years;
* Under the condition of bilateral cycloplegic autorefraction, the spherical refractive error of -6.00 to -0.50 D in each eye and astigmatism of not more than 1.50 D and anisometropia of not more than 1.50 D;
* Best-corrected visual acuity of equal or better than 0.00 LogMAR (>= 1.0 as Snellen).
* The intraocular pressure of 10 to 21mmHg.
* Volunteer to participate in this clinical trial with signature of the informed consent form.

Exclusion Criteria:

* History of eye injury or intraocular surgery;
* Clinically abnormal slit-lamp findings
* Abnormal fundus examination
* Ocular disease, such as uveitis and other inflammatory diseases, glaucoma, cataract, fundus diseases, eye tumors, dominant strabismus, and any eye diseases that affect visual function;
* Systemic diseases causing low immunity (such as diabetes, Down's syndrome, rheumatoid arthritis, psychotic patients or other diseases that researchers think are not suitable for wearing glasses);
* Participation of the drug clinical trial within three month and the device clinical trial within one month;
* Only one eye meets the inclusion criteria;
* Unable to have regular follow-up
* Participation of any myopia control clinical research trial within three months, and currently using rigid contact lenses (including nursingproducts), multifocal contact lenses, progressive multifocal lenses and other specially designed myopia control lenses, atropine drugs, etc.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes of spherical equivalent refraction (SER) at two years | 2 years
  The difference of SER (Diopter) at two years compared with baseline SER. SER will be measured after cycloplegia.

SECONDARY OUTCOMES:
Changes of axial length (AL) at two years | 2 years
  The difference of AL (mm) at two years compared with baseline AL. AL will be measured by IOLMaster-700.
Visual scale score at two years | 2 years
  Visual scale score measured by the Chinese version of the pediatric refractive error profile2 (PREP2) is scaled from 0 (poor quality of life) to 100 (good quality of life).
Incidence of adverse event during study period | 2 years
  Adverse event is a comprehensive qualitative outcome measure that will be evaluated based on the participants' symptoms and signs, intraocular pressure, slit lamp and fundus examinations, as well as lens and frame damage. The evaluation will be conducted every six months according to the predetermined definition of abnormalities in the above examinations.

OTHER OUTCOMES:
Change of lens thickness (LT) at two years | 2 years
  The difference of LT (mm) at two years compared with baseline LT. LT will be measured by IOLMaster-700.
Change of corneal power (CP) at two years | 2 years
  The difference of CP (diopter) at two years compared with baseline CP. CP will be measured by IOLMaster-700.
Best corrected visual acuity at two years | 2 years
  Best corrected visual acuity will be measured at baseline and two years by EDTRS visual acuity chart.
Binocular visual function at two years | 2 years
  Binocular visual function which is a qualitative outcome assessed by a series of tests will be measured every half year.
Change of choroidal thickness at two years | 2 years
  The difference of Choroidal thickness (μm) at two years compared with baseline measure. Choroidal thickness will be measured by OCTA.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Ge, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China